CLINICAL TRIAL: NCT04960787
Title: A Randomized Trial Addressing Cancer-Related Financial Hardship Through Delivery of a Proactive Financial Navigation Intervention (CREDIT)
Brief Title: Financial Navigation Program to Improve Understanding and Management of Financial Aspects of Cancer Care for Patients and Their Spouses
Acronym: CREDIT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: S1912CD; NCI-2021-00579 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1912CD (Other: SWOG); SWOG-S1912CD (Other: DCP); S1912CD (Other: CTEP); R01CA248656 (NIH); UG1CA189974 (NIH)
Record Dates: First submitted 2021-06-08; First posted 2021-07-14 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Metastatic Malignant Solid Neoplasm; Recurrent Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasm Metastasis | interventions — Early Intervention, Educational; Educational Status; Methods; Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (usual care) (Active Comparator): Patients receive financial literacy training consisting of watching online educational videos over 2-8 minutes. Patients also complete questionnaires over 30-60 minutes about education, employment, finances (assets, debt), insurance, and quality of life (financial worry) and have credit reports assessed at baseline and 3, 6, and 12 months.
  If participating, spouse/partner caregivers will receive the same intervention, and will complete questionnaires and have credit reports assessed at baseline and 3, 6, and 12 months.
  Interventions: Other: Educational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (financial navigation intervention) (Experimental): Patients receive financial literacy training consisting of watching online educational videos over 2-8 minutes. Patients also meet with CENTS counselor and PAF case manager over approximately 1 hour every month for 6 months (with each group). Patients also complete questionnaires over 30-60 minutes about education, employment, finances (assets, debt), insurance, and quality of life (financial worry) and have credit reports assessed at baseline and 3, 6, and 12 months.
  If participating, spouse/partner caregivers will receive the same intervention, and will complete questionnaires and have credit reports assessed at baseline and 3, 6, and 12 months.
  Interventions: Other: Educational Intervention; Behavioral: Patient Navigation; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Watch online educational videos
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Behavioral: Patient Navigation — Meet with CENTS counselor and PAF case manager
  Other Names: Patient Navigator Program
  Arms: Group II (financial navigation intervention)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This clinical trial examines a financial navigation program in helping patients (and their spouses or partner caregivers, if participating) understand and better manage the financial aspects of cancer care. Cancer patients and their spouse/partner caregivers may be at high risk for financial problems because of the cost of cancer treatment. A financial navigator is a person or team who works with patients and their families to help them reduce stress or hardship related to the cost of cancer treatment. Financial navigators help patients understand their out-of-pocket expenses and what their health insurance plans may cover. Financial navigation may also help patients set up payment plans, find cost-saving methods for treatments, and improve access to healthcare services that the patient needs. Providing financial navigation to patients may help reduce financial worries and improve quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether a proactive financial navigation program for patients planning to receive anti-cancer treatment decreases the risk of material household financial hardship over 12 months among patients with newly diagnosed or recurrent metastatic solid tumor, or a newly diagnosed hematologic malignancy.

SECONDARY OBJECTIVES:

I. To examine whether proactive financial navigation improves patient quality of life.

II. To examine whether proactive financial navigation decreases financial worry among patients relative to usual care and explore the extent to which financial worry correlates with financial hardship.

III. To explore whether the proactive financial navigation intervention leads to decreased cost-related medication non-adherence and fewer patient emergency department (ED) visits and unplanned hospital admissions.

ADDITIONAL OBJECTIVES:

I. To explore the impact of proactive financial navigation on spouse/partner caregiver financial hardship, quality of life, and caregiver burden and evaluate the concordance between patient and caregiver credit data.

II. To explore the utilization of financial navigation services by younger, financially fragile, and lower income patients and households and evaluate the moderator effect of age, financial fragility, and income on the impact of the proactive financial navigation intervention.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive financial literacy training consisting of watching online educational videos over 2-8 minutes. Patients also complete questionnaires over 30-60 minutes about education, employment, finances (assets, debt), insurance, and quality of life (financial worry) and have credit reports assessed at baseline and 3, 6, and 12 months.

GROUP II: Patients receive financial literacy training consisting of watching online educational videos over 2-8 minutes. Patients also meet with Consumer Education and Training Services (CENTS) counselor and Patient Advocate Foundation (PAF) case manager over approximately 1 hour every month for 6 months (with each group). Patients also complete questionnaires over 30-60 minutes about education, employment, finances (assets, debt), insurance, and quality of life (financial worry) and have credit reports assessed at baseline and 3, 6, and 12 months.

Spouse/partner caregiver participation is optional. If a spouse/partner caregiver is participating in the trial along with the patient. If participating, the spouse/partner caregiver receives the same intervention as the patient and will complete questionnaires and have credit reports assessed at baseline and 3, 6, and 12 months.

SAMPLE SIZE: Study participants include both patients and optional spouse/partner caregivers. Study enrollment targets are based entirely on patients, but the anticipated number of participants includes both groups. We expect to enroll 326 patients and approximately 196 spouse/partner caregivers for a total of 522 anticipated participants, but the study will be closed to accrual when the patient accrual target of 326 is reached, regardless of the number of participating spouse/partner caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of a metastatic solid tumor or a hematologic malignancy and must receive anti-cancer treatment (i.e. chemotherapy, hormonal therapy, targeted therapy, biologic therapy, immune therapy, bone marrow transplant). Registration must occur within 180 days after diagnosis of metastatic or stage IV solid tumor or treatment-requiring hematologic malignancy. Patients with indolent hematologic diseases undergoing observation alone are not eligible; patients with previously diagnosed hematologic cancers progressed to the point of requiring systemic therapy are eligible, so long as the progression occurred within the previous 180 days. Biopsy confirmation of metastatic disease is not required
* Patients with recurrent solid tumors will be allowed as long as 1) this is the first presentation of metastatic disease and 2) the diagnosis of the metastasis is at least 180 days (6 months) after the diagnosis date of the previous earlier stage cancer
* Patients with a history of secondary malignancy are allowed as long as they were not diagnosed within the previous 24 months, are not on active therapy, and are disease-free. Patients with adequately treated basal cell or squamous cell skin cancer, and in situ cervical cancer at any point prior to enrollment are eligible
* Patients who have started anti-cancer treatment for the current diagnosis must have started within 90 days prior to registration
* Patients who are planning to start anti-cancer treatment for the current diagnosis must start within (=<) 30 days after registration
* Patients are allowed to be co-enrolled on other clinical trials (including non-treatment studies and studies that may or may not include investigational drugs)
* Patients must be at least 18 years of age
* Patients must have a Zubrod performance status of 0-2
* Patients must complete the baseline patient reported outcomes (PRO) questionnaires prior to registration and must be able to complete questionnaires in English or Spanish
* Patients must provide their full name, primary address in the United States (U.S.), birth date and social security number at registration for the purposes of accessing credit report data. (This may be obtained directly from the patient, study questionnaires, or the medical record)
* Patients must provide email and/or telephone number for the purposes of being contacted by financial navigators Spouse/partner caregiver participation is optional.
* Spouse/partner caregiver must be living in the same household as the eligible patient and be either legally married, in a common law marriage, or be an intimate partner/significant other of the participant*
* Spouse/partner caregivers must be at least 18 years of age
* Spouse/partner caregivers must provide their full name, primary address in the U.S., birth date and social security number at registration for the purposes of accessing credit report data
* Spouse/partner caregivers must provide email and/or telephone number for the purposes of being contacted by the financial navigators
* Spouse/partner caregivers must be able to complete questionnaires in English or Spanish and must complete the baseline questionnaires prior to patient registration

  *The study team acknowledges that other types of caregivers may also face financial hardship following a patient's cancer diagnosis and may similarly benefit from financial education and navigation. The decision to focus solely on spouse or partner caregivers was scientific, to understand how caregivers who share household finances experience financial hardship.
* Participants (patients and caregivers, when participating) must sign and give written informed consent in accordance with institutional and federal guidelines. Use of legally-authorized representative is not permissible for this study. Documentation of informed consent via remote consent is permissible
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Exclusion Criteria:

* Patients may not be enrolled in hospice care at the time of registration
* Non-spouse/partner caregivers such as friends, adult children, parents, or other relatives living in the same household as the patient are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Patient financial hardship | Up to 12 months
  Defined as one or more of the following: from the patient's credit report within 12 months: any new loans (bank or home equity); exhausting lines of credit by reaching limits on credit cards and home equity loans; credit or other payment delinquencies; becoming subject to a lien, judgment, or other collection process; personal bankruptcy filings. Will conduct a multivariable logistic regression (outcome = patient financial hardship; independent variable = intervention versus [vs.] control), adjusting for demographic, clinical, financial and practice characteristics.

SECONDARY OUTCOMES:
Quality of life: patient | Up to 12 months
  As measured by composite European Quality of Life Five Dimension Five Level Scale (EQ-5D-5L). The proportion of patients in each arm who experience improved, unchanged, or worsened EQ-5D scores from baseline to 3, 6 (and 12) months will be compared using Fisher's exact test. Mean score changes will be compared using two group t tests. A multivariate linear regression model, with worsening score as the dependent variable and study arm as the independent variable will be performed.
Financial worry | Up to 12 months
  Will be measured by the Comprehensive Score for Financial Toxicity-Patient Reported Outcome Measure (COST-Functional Assessment of Chronic Illness Therapy [FACIT] version 2; Financial Toxicity Scale ranges from 0-44, with higher scores indicating greater financial well-being). Mean scores (and standard deviation [SD]) at 3, 6 and 12 months will be compared between intervention and usual care patients using two sample t tests.
Treatment adherence: Number of patients | Up to 12 months
  Number of patients by study arm self-reporting that they did or did not skip medication doses or refuse/decline recommended therapy due to cost concerns.
Treatment adherence: Proportion of patients | Up to 12 months
  Proportion of patients by study arm self-reporting that they did or did not skip medication doses or refuse/decline recommended therapy due to cost concerns.
Emergency department/hospital use | Up to 12 months
  Will be abstracted from patients' medical records by site staff. Investigators will categorize visits as anticipated (for chemotherapy or planned procedures) versus unanticipated (complication or treatment side-effect). The cumulative incidence of emergency department and unanticipated hospital use will be calculated by arm to account for death as a competing risk and compared using Cox regression, adjusting for covariates.

OTHER OUTCOMES:
Spouse/partner caregiver financial hardship | Up to 12 months
  Defined as one or more of the following: from the spouse/partner caregiver's credit report within 12 months: any new loans (bank or home equity); exhausting lines of credit by reaching limits on credit cards and home equity loans; credit or other payment delinquencies; becoming subject to a lien, judgment, or other collection process; personal bankruptcy filings. Will conduct a multivariable logistic regression (outcome = spouse/partner financial hardship; independent variable = intervention versus [vs.] control), adjusting for demographic, clinical, financial and practice characteristics.
Spouse/partner caregiver burden | Up to 12 months
  As measured by the social well-being (Social Concerns, range:0-90, higher scores better) subscale of the City of Hope Quality of Life Family questionnaire. Mean score changes will be compared using two group t tests. A multivariate linear regression model, with worsening score as the dependent variable and study arm as the independent variable will be performed.
Quality of life: spouse/partner caregiver | Up to 12 months
  As measured by City of Hope Quality of Life Family subscale scores (Physical Well Being (0-50), Psychological Well Being (0-110); higher scores better). We will determine the proportion of spouse/partner caregivers in each arm who experience improved, unchanged, or worsened Quality of Life Family scores (composite scores for physical, psychological, and social well-being subscales) from baseline to 3, 6 (and 12) months and compare using Fisher's exact test. Mean score changes will be compared using two group t tests. A multivariate linear regression model, with worsening score as the dependent variable and study arm as the independent variable will be performed.
Community/clinic assistance | Up to 12 months
  Control arm dyads will be surveyed about availability (or lack), access to, and use of financial assistance via their treating clinic or community-based resources.
Qualitative assessment of the intervention | Up to 12 months
  Qualitative Assessment of the Intervention: Intervention arm dyads will be surveyed about availability and use of financial assistance and navigation services with Consumer Education and Training Services (CENTS) and/or Patient Advocate Foundation (PAF). CENTS and PAF will document all interactions with the intervention dyads and specific details about all counseling, assistance, and interventions provided for the dyad over the 6-month intervention period using Medidata Rave.

CONTACTS AND LOCATIONS:
Overall Officials: Veena Shankaran, Principal Investigator — SWOG Cancer Research Network
Locations (266):
- United States (264):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Epic Care-Dublin, Dublin, California
  - Kaiser Permanente Dublin, Dublin, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Beebe South Coastal Health Campus, Frankford, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Augusta University Medical Center, Augusta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Bromenn Lifecare Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed University of Kansas Health System, Hays, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates, Baton Rouge, Louisiana
  - Our Lady of the Lake Medical Oncology, Baton Rouge, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Stephens Memorial Hospital, Norway, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Maine Medical Partners - South Portland, South Portland, Maine
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Hackettstown Medical Center, Hackettstown, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Newton Medical Center, Newton, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Lovelace Radiation Oncology, Albuquerque, New Mexico
  - Lovelace Women's Hospital, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Lourdes Hospital, Binghamton, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Kaiser Permanente Northwest, Portland, Oregon
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Waccamaw Oncology - Georgetown, Georgetown, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Waccamaw Oncology-Murrells Inlet, Murrells Inlet, South Carolina
  - Waccamaw Oncology-Myrtle Beach, Myrtle Beach, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Wellmont Medical Associates-Bristol, Bristol, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Valley Medical Center, Renton, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
- Puerto Rico (2):
  - Doctors Cancer Center, Manatí
  - Centro Comprensivo de Cancer de UPR, San Juan